CLINICAL TRIAL: NCT02742298
Title: Electrical Impedance Myography and Muscle Ultrasound: Longitudinal Measures in Pompe Disease
Brief Title: Pompe Disease QMUS and EIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: Pro00072199
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-02

CONDITIONS: Pompe Disease
Keywords: Neuromuscular Ultrasound; Electrical Impedance Myography
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QMUS (Other): All patients will undergo serial quantitative muscle ultrasound.
  Interventions: Device: Muscle ultrasound
- EIM (Other): All patients will undergo serial electrical impedance myography measures.
  Interventions: Other: Electrical Impedance Myography

INTERVENTIONS:
Device: Muscle ultrasound — Ultrasound images of limb muscles will be collected.
  Arms: QMUS
Other: Electrical Impedance Myography — A painless current passes through the skin and surface electrodes are used to record the impedance through muscle.
  Arms: EIM

SUMMARY:
Study Objectives:

1. Determine the correlation between quantitative muscle ultrasound (QMUS), electrical impedance myography (EIM) and currently accepted measures of physical function.
2. Determine the reliability of EIM measures performed in the home through use of a hand held device.
3. Determine if QMUS and EIM can detect pre-clinical changes in Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Pompe disease.

Exclusion Criteria:

* Age <18 years
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Percent change in muscle ultrasound echointensity as compared to baseline | Baseline, 1-2 years
Percent change in muscle electrical impedance myography as compared to baseline | Baseline, 1-2 years

SECONDARY OUTCOMES:
Inter-rater reliability of muscle ultrasound and electrical impedance myography measures | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Hobson-Webb, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No